CLINICAL TRIAL: NCT05987501
Title: Prospective Study to Evaluate the Role of Contrast-enhanced Ultrasound (CEUS) and Elastography in Predicting Clinical and Endoscopic Remission (Deep Remission) in Inflammatory Bowel Disease
Brief Title: Multimodal Ultrasound in Inflammatory Bowel Diseases
Acronym: CELESTIAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zocco Maria Assunta, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2743
Record Dates: First submitted 2023-03-16; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): patients with Crohn's disease or Ulcerative Colitis needing to begin biologic treatment
  Interventions: Diagnostic Test: Multimodal ultrasound

INTERVENTIONS:
Diagnostic Test: Multimodal ultrasound — Contrast enhanced ultrasound and shear wave elastography on target intestinal loop are perfomed before and at different timepoints after treatment induction

SUMMARY:
The role of intestinal ultrasound in treatment monitoring has recently gained increasing interest thanks to its non-invasiveness, cost-effectiveness and largely availability. Moreover, new ultrasonographic tools, particularly dynamic contrast-enhanced ultrasound (D-CEUS) and shear wave elastography (SWE) can provide further useful information, such as a quantitative estimation of bowel intramural microvacularization and tissue stiffness.

Aim of this study is to evaluate the role of D-CEUS and SWE in predicting deep remission at 12 months from treatment induction in IBD.

DETAILED DESCRIPTION:
Background: Clinical remission is no more considered an appropriate therapeutic target for Inflammatory Bowel Diseases (IBD) and other parameters such as endoscopic and transmural remission are now recognized as prognostic factors ("deep remission"). Correctly monitoring treatment response is crucial to rapidly adequate therapeutic algorithms avoiding complications. The role of intestinal ultrasound in treatment monitoring has recently gained increasing interest thanks to its non-invasiveness, cost-effectiveness and largely availability. Moreover, new ultrasonographic tools, particularly dynamic contrast-enhanced ultrasound (D-CEUS) and shear wave elastography (SWE) can provide further useful information, such as a quantitative estimation of bowel intramural microvacularization and tissue stiffness.

Primary objective: to evaluate the role of D-CEUS and SWE in predicting deep remission at 12 months from treatment induction in IBD.

Secondary objectives:

* To evaluate the relationship between clinical activity and CEUS/elastography parameters
* To evaluate the relationship between endoscopic activity and CEUS/elastography parameters
* To evaluate the relationship between inflammation indices and CEUS/elastography

Exploratory aims:

* To evaluate the relationship between CEUS/elastography parameters and serum biomarkers of fibrosis
* To evaluate the relationship between CEUS/elastography parameters and faecal microbiota in a subset of patients Study design: Prospective, interventional, single-center study. Methods: 50 consecutive patients with Crohn's disease or Ulcerative Colitis needing to begin biologic treatment according to international guidelines and with an affected intestinal segment detectable in B-mode ultrasound will be enrolled in the Unit of Internal Medicine and Gastroenterology of the Policlinico Gemelli. Exclusion criteria will be induction of biologic therapy in prophylaxis after surgery in Crohn's disease, lack of visualization of affected intestinal tract (eg. obesity), diagnosis of undetermined colitis, hearth failure, known allergy to ultrasound contrast agents, pregnancy and lactation. Colonoscopies, blood tests and ultrasound evaluations (B-mode ultrasound, elastography and CEUS) will be performed as per normal clinical practice. Data obtained from these procedures will be recorded and analyzed specifically for the study. The only study-specific procedures are the collection of fecal samples for microbiota evaluation, urine samples for metabolomics evaluation and an additional blood sample for evaluation of fibrosis biomarkers, both collected at the time of recruitment. The additional blood sample will be taken from the same peripheral venous access route used for blood sampling in normal clinical practice. Ileal elastography and CEUS will be performed before starting treatment and after 2/3, 8 and 16 weeks, 6 months, 12 months, 24 months and 36 months. If indicated by clinical assessment, some patients will be re-evaluated after 3 weeks. Clinical assessment will include Harvey-Bradshaw index or Mayo score, blood cell count, CRP and ESR, as per clinical practice. An additional blood sampling will be done for fibrosis biomarker evaluation. In particular, we will do multiple analysis (Bio-Plex, Biorad ) for IL-1ra, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12, IL-13, IL-15, IL-17, Eotaxin, basic FGF, G-CSF, GM-CSF, IFN-g, IP-10, MCP-1, MIP-1a, PDGF-bb, MIP-1b, RANTES, TNF-a, VEGF, TL -1a, TGF-b, IL-33, ST2. Data about the clinical outcome (i.e. surgery, hospitalizations, need for steroids…) and biomarkers of fibrosis will be collected up to 36 months after the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* diagnosis of Crohn's disease or Ulcerative Colitis
* indication to start biologic treatment according to international guidelines
* affected intestinal segment detectable in B-mode ultrasound

Exclusion Criteria:

* induction of biologic therapy in prophylaxis after surgery in Crohn's disease
* lack of visualization of affected intestinal tract (eg. obesity)
* diagnosis of undetermined colitis
* hearth failure
* known allergy to ultrasound contrast agents
* pregnancy
* lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
predicting treatment response | 12 months after treatment induction
  to quantify peak enhancement intensity in Arbitray Units AU (measured by analysing D-CEUS time-intensity curves) in patients with inflammatory bowel diseases undergoing biological treatment, stratified according to 12-months response to treatment (responders vs non-responders)

SECONDARY OUTCOMES:
predicting treatment response | 12 months after treatment induction
  to quantify the other D-CEUS parameters (measured by analysing D-CEUS time-intensity curves) in patients with inflammatory bowel diseases undergoing biological treatment, stratified according to 12-months response to treatment (responders vs non-responders)
predicting treatment response | 12 months after treatment induction
  to quantify mean intestinal loop stiffness (measured by shear wave elastography) in patients with inflammatory bowel diseases undergoing biological treatment, stratified according to 12-months response to treatment (responders vs non-responders)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

REFERENCES:
- [Derived] Ainora ME, Liguori A, Mignini I, Cintoni M, Galasso L, Laterza L, Lopetuso LR, Garcovich M, Riccardi L, Gasbarrini A, Scaldaferri F, Zocco MA. Multimodal dynamic ultrasound approach as predictor of response in patients with Crohn's disease treated with ustekinumab. Therap Adv Gastroenterol. 2024 Jun 22;17:17562848241259289. doi: 10.1177/17562848241259289. eCollection 2024. PMID 38912296